CLINICAL TRIAL: NCT02881242
Title: A Single-Arm, Open-Label, Two-Stage Phase II Study of the MEK 1/2 Inhibitor Trametinib in Men With Progressive Metastatic Castrate Resistant Prostate Cancer
Brief Title: Trametinib in Treating Patients With Progressive Metastatic Hormone-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Stand Up To Cancer (Other); Novartis (Industry); Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-001044; NCI-2016-01201 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Prostate Carcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (trametinib) (Experimental): Patients receive trametinib PO QD. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Trametinib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist

SUMMARY:
This phase II trial studies how well trametinib works in treating patients with hormone-resistant prostate cancer that is growing or getting worse and has spread to other parts of the body. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. To assess the activity of trametinib in metastatic castration resistant prostate cancer (mCRPC) that has progressed on either enzalutamide or abiraterone acetate.

SECONDARY OBJECTIVES I. Durability of prostate specific antigen (PSA) response as measured by the time to PSA progression as defined by Prostate Cancer Working Group 2 guidelines for PSA progression.

II. Maximal PSA response. III. Quality of life by Functional Assessment of Cancer Therapy- Prostate (FACT-P).

IV. Time to initiation of alternative antineoplastic therapy. V. Time to radiographic progression. VI. Objective response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines.

VII. Overall survival measured as time from enrollment until death. VIII. Safety and tolerability. IX. Analysis of trametinib target engagement of mitogen-activated extracellular signal-related kinase (MEK1/2) is assessed by presence of p-ERK, the primary phosphorylation target of activated MEK1/2, in pre-treatment and at progression radiographically directed metastatic tumor biopsies by immunohistochemistry evaluation of p-ERK. Markers of cell proliferation (Ki67) and apoptosis (p27) will also be assessed.

XI. Investigation of molecular correlates to resistance and sensitivity to trametinib using pre-treatment and at progression metastatic biopsies.

XII. Discovery of one or a set of possible discriminative networks that are associated with a response to trametinib.

XII. Enrichment for patients in the second phase who have tumors exhibiting genomic features associated with a response to trametinib.

XIV. Analyses of circulating tumor deoxyribonucleic acid (ctDNA) for genomic aberrations correlated to treatment response.

OUTLINE:

Patients receive trametinib orally (PO) once daily (QD). Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2 and 4 weeks, and then every 4 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* Histologically confirmed prostate cancer (not exclusive of adenocarcinoma)
* mCRPC that has progressed on at least 1 therapy progression (defined as Prostate Cancer Working Group 2 [PCWG2] or at investigators' discretion) approved for treatment of mCRPC, one of which must include abiraterone acetate and/or enzalutamide
* Metastatic tumor that has been biopsied
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Willing to undergo biopsy of a metastatic lesion at the time of progression
* Patients must have ongoing therapy to maintain serum testosterone < 50 ng/dL
* Absolute neutrophil count > 1,500/uL during screening evaluation
* Platelet count > 100,000/uL during screening evaluation
* Hemoglobin > 9 g/dL during screening evaluation
* Total bilirubin within the reference range during screening evaluation
* Alanine aminotransferase (ALT) within the reference range during screening evaluation
* Aspartate aminotransferase (AST) within the reference range during screening evaluation
* Creatinine < (1.5 mg/dL) during screening evaluation (> 1.5 is allowed if epidermal growth factor receptor [EGFR] > 45 mL/min/1.73 m^2)
* International normalized ratio (INR) < 1.3 (or < 3 if on warfarin or other anticoagulants) during screening evaluation
* Left ventricular ejection fraction (LVEF) >= 45% as measured by echocardiogram during screening evaluation
* Electrocardiogram (EKG) without clinically significant abnormality

Exclusion Criteria:

* A history of retinal vein occlusion (RVO) or risks factors for RVO
* A history of retinal pigment epithelial detachment (RPED) or risk factors for RPED
* Clinically significant abnormality on ophthalmologic examination during screening evaluation
* Clinically significant cardiovascular disease including:

  * LVEF < 45% measured by echocardiogram
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months
  * Uncontrolled angina within 3 months
  * New York Heart Association (NYHA) class III or IV congestive heart failure
  * Clinically significant abnormality on EKG
  * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)
  * Patients with intra-cardiac defibrillators or permanent pacemakers
* Presence of a comorbid disease or medical condition that would impair the ability of the patient to receive or comply with the study protocol
* History of interstitial lung disease or pneumonitis
* Use of any medication or herbal products that may have hormonal anti-prostate cancer activity and/or are known to modulate PSA levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone per day within 4 weeks of enrollment
* Prior use of trametinib or other mitogen activated protein kinase (MAPK) inhibitor in any context
* Known or suspected brain metastasis or active leptomeningeal disease or spinal cord compression
* Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within last 3 months, inflammatory bowel disease)
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 30 days of enrollment and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days of enrollment
* Hospitalization within 30 days of enrollment for cancer related events
* History of another malignancy within the previous 5 years other than curatively treated non-melanoma skin cancer
* Use of an investigational agent within 4 weeks of enrollment
* Use of any medications known to affect the serum androgen level
* Any condition or reason that, in the opinion of the investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
PSA response rate | At 12 weeks
Response rate assessed by RECIST criteria | Up to 24 weeks
  Will be defined as decline in PSA of 30% or more, any decline of PSA of 50% or more, partial or complete response at 12 weeks, and freedom from radiographic progression at 24 weeks.

SECONDARY OUTCOMES:
Change in markers of cell proliferation (Ki67) and apoptosis (p27), assessed by immunohistochemistry | Baseline up to 24 weeks
  Mixed effects logistic regression models to assess changes in markers over time, correlations between markers over time and associations between markers and treatment response (conditional logistic regression) will be used.
Change in trametinib target engagement of MEK1/2 defined by the presence of p-ERK, assessed by immunohistochemistry | Baseline up to 24 weeks
  Mixed effects logistic regression models to assess changes in markers over time, correlations between markers over time and associations between markers and treatment response (conditional logistic regression) will be used.
Durability of PSA response as measured by time to PSA progression as defined by PCWG2 guidelines | Up to 30 months
Incidence of adverse events, graded according to the Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 months
Maximal PSA response | Up to 30 months
Molecular correlates defined by gene expression, assessed using ribonucleic acid-sequencing, and mutational events, assessed using DNA exome-seq | Up to 24 weeks
  Statistical bootstrap and Pearsons Correlation will be used to determine the relationship of phenotype to mutations and clinical variables. Fisher exact tests and logistic regression models will be used to evaluate the relationships between specific variations and treatment response.
Objective radiographic response rate according to RECIST guidelines | Up to 24 weeks
Overall survival | Time from enrollment until death, assessed for up to 30 months
Quality of life, assessed by FACT-P | Up to 30 months
Time to initiation of alternative anti-neoplastic therapy | Up to 30 months
Time to radiographic progression | Up to 24 weeks

OTHER OUTCOMES:
ctDNA genomic aberrations, assessed by exome sequencing | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Rettig, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States